CLINICAL TRIAL: NCT04312373
Title: Efficacity of a Rigid Ankle Foot Orthosis for Persons With Ankle Osteoarthritis
Acronym: SCED-SA
Status: Completed | Type: Observational
Sponsor: Union de Gestion des Etablissements des Caisses d'Assurance Maladie - Nord Est (Other)
Responsible Party: Sponsor
Other Study IDs: IRR-2018-SCED
Record Dates: First submitted 2020-02-27; First posted 2020-03-18 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Ankle Osteoarthritis
Keywords: Ankle Osteoarthritis; Ankle Foot Orthosis; Ankle Arthrodesis; Single Case Experimental Design

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Ankle Foot Orthosis — According to the SCED methodology, patients were fitted with ankle foot orthosis intermittently, during 4 phases, in the following order : without orthosis (A1), with orthosis (B1), again without orthosis (A2) and again with orthosis (B2).
  All the phases were carried out over one day.

SUMMARY:
Ankle osteoarthritis (AOA) is a typical long-term complication of an ankle injury. Pain during walking is the main symptom that limits walking distance. Non-surgical treatments could be used to decrease pain. The gold standard treatment for end-stage OA is definitive surgical ankle arthrodesis.

The purpose of this study was to assess the effectiveness of a rigid ankle-foot orthosis (R-AFO) for walking pain in a population suffering from AOA.

DETAILED DESCRIPTION:
This study used the SCED introduction/withdrawal methodology to assess the efficacy of R-AFO on pain and walking distance in the 2-minute walk test (2MWT). Each patient is his or her own comparator. During phase A, considered as the baseline, the patient performs the 2MWT without R-AFO. During phases B, considered as the introduction phases, the patient performs the tests with R-AFO. These tests are performed repeatedly and at regular intervals. The time of transition between phases has been randomized to have a minimum of 3 trials per phase.

At the end of each test, an visual analogue scale for the pain and the walking distance travelled during the 2MWT were recorded.

ELIGIBILITY:
Inclusion Criteria:

* primary or post-traumatic one-sided Ankle osteoarthritis (AOA)
* Able to walk at least two minutes

Exclusion Criteria:

* cardiovascular diseases
* respiratory diseases that prevent subjects from performing the walking tests
* neurologic or orthopaedic diseases which could affect their gait (excluding AOA)
* inability to understand study instructions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from AOA
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
Evolution of the distance travelled during the 2MWT between each phase | 1 day, starting from the baseline
  In m.
Evolution of the Visual Analogue Scale (VAS) for walking ankle pain between each phase | The VAS was performed after each 2MWT. All 2MWT were completed in one day.
  Scale from 0 to 10, the higher the score the higher the pain.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Paysant, PhD-MD, Study Chair — Institut Régional de Médecine Physique et de Réadaptation
Locations (1):
- Institut Régional de Médecine Physique et de Réadaptation, Nancy, France